CLINICAL TRIAL: NCT04576871
Title: Pilot Study of PSMA-TRT Re-treatment Utilizing 225Ac-J591
Brief Title: Re-treatment 225Ac-J591 for mCRPC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-01021286
Record Dates: First submitted 2020-09-24; First posted 2020-10-06 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heavily Exposed (Experimental)
  Interventions: Drug: 225Ac-J591
- Moderately Exposed (Experimental)
  Interventions: Drug: 225Ac-J591

INTERVENTIONS:
Drug: 225Ac-J591 — In this study, subject enrollment will be done in a re-treatment design. A single dose of 225Ac-J591 given at the specified dose per cohort. The initial planned dose level will be determined based upon prior radioactivity exposure level. Those with moderate exposure (up to 30 GBq of 177Lu) will start with 65 KBq/Kg and those with heavy prior exposure (more than 30 Gbq of 177Lu or any 225Ac) will start with 50 KBq/Kg.
  Other Names: 68Ga-PSMA-HBED-CC injection for PET/CT Scan at screening, week 12 and week 24

SUMMARY:
The purpose of this study is to find out if re-treatment with 225Ac-J591 can be given without severe side effects.

DETAILED DESCRIPTION:
This is an open-label, pilot study designed to determine the safety of PSMA-TRT re-treatment with 225Ac-J591, which will be given in a single dose on D1, in men with progressive mCRPC. If the patient responds and tolerates this dose, another may be given upon progression, provided at least 12 weeks after the initial dose.

This research study is being done because the standard treatments for prostate cancer that has spread beyond the prostate gland are intended to minimize the adverse effects of the disease and make men live longer. These treatments, however, are not curative so additional treatments are needed. Prostate-specific membrane antigen (PSMA) is a protein that is on the surface of most prostate cancer cells. It is absent from most other normal places in the body, but is present to some degree in the kidney, small intestine, salivary glands, and brain. J591 is a monoclonal antibody (an engineered protein) which recognizes PSMA. Actinium-225 (225Ac) is a small radioactive particle that emits alpha-particles (damaging/ionizing radiation). 225Ac-J591 is the combination compound that has the radioactive particle linked to J591. It is designed so that J591 will recognize PSMA and drags the radioactive particle 225Ac with it wherever it goes. This drug used currently is not FDA approved for any indication and is considered experimental.

In the first part of the study, a small group of subjects will receive a dose of 225Ac-J591 based upon a prior study. If that dose does not lead to severe side effects in many subjects, an additional small group will be treated. If the initial dose leads to too many severe side effects, another group will receive a lower dose. If it is determined by a physician that a subject's tumor has responded favorably to treatment, did not experience severe side effects and subject in agreement, then the subject will be allowed to receive one additional dose of the study drug 225Ac-J591, provided that at least 3 months have passed since the initial dose. For subjects receiving re-treatment, they will also participate in the same study procedures and followed for treatment including short-term and long-term follow up.

All treatment visits and all visits involving investigational PSMA PET imaging are required to be performed at the Weill Cornell Medicine - NewYork Presbyterian site located in the upper east side of Manhattan.

ELIGIBILITY:
Inclusion Criteria

1. Histologically or cytologically confirmed adenocarcinoma of prostate
2. Documented progressive metastatic CRPC based on Prostate Cancer Working Group 3 (PCWG3) criteria, which includes at least one of the following criteria:

   * PSA progression
   * Objective radiographic progression in soft tissue
   * New bone lesions
3. ECOG performance status of 0-2
4. Have serum testosterone ≤ 50 ng/dL. Subjects must continue primary androgen deprivation with an LHRH/GnRH analogue (agonist/antagonist) if they have not undergone orchiectomy
5. Have previously been treated with at least one of the following in any disease state:

   * Androgen receptor signaling inhibitor (such as enzalutamide)
   * CYP 17 inhibitor (such as abiraterone acetate)
6. Have previously received taxane chemotherapy (in any disease state), been determined to be ineligible for taxane chemotherapy by their physician, or refused taxane chemotherapy
7. Age ≥ 18 years
8. Patients must have normal organ and marrow function as defined below:

   * Absolute neutrophil count: ≥ 2,000 cells/mm3
   * Hemoglobin: ≥9 g/dL
   * Platelet count: ≥150 x 10^3/ microliter
   * Serum creatinine: ≤1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/min/1.73 m^2 by Cockcroft-Gault
   * Serum total bilirubin: ≤1.5 x ULN (unless due to Gilbert's Syndrome in which case direct bilirubin must be normal)
   * Serum AST and ALT ≤3 x ULN in absence of liver metastases; < 5x ULN if due to liver metastases (in both circumstances bilirubin must meet entry criteria)
9. Ability to understand and the willingness to sign a written informed consent document
10. In the opinion of the investigator, history of clinical benefit with treatment using PSMA-TRT and no dose-limiting toxicity. Clinical benefit might be assessed by PSA changes, CTC changes, radiographic changes, and/or symptomatic improvement

Exclusion Criteria

1. Implantation of investigational medical device ≤4 weeks of Treatment Visit 1 (Day 1) or current enrollment in oncologic investigational drug or device study
2. Use of investigational drugs ≤4 weeks or <5 half-lives of Cycle 1, Day 1 or current enrollment in investigational oncology drug or device study
3. Prior systemic bone-seeking beta-emitting radioisotopes. Prior radium-223 is allowed provided last dose was at least 12 weeks prior to C1D1 on this protocol
4. History of deep vein thrombosis and/or pulmonary embolus within 1 month of C1D1
5. Other serious illness(es) involving the cardiac, respiratory, CNS, renal, hepatic or hematological organ systems which might preclude completion of this study or interfere with determination of causality of any adverse effects experienced in this study
6. Radiation therapy ≤4 weeks of Day 1 Cycle 1
7. Having partners of childbearing potential and not willing to use a method of birth control deemed acceptable by the principle investigator and chairperson during the study and for 1 month after last study drug administration
8. Currently active other malignancy other than non-melanoma skin cancer. Patients are considered not to have "currently active" malignancy if they have completed any necessary therapy and are considered by their physician to be at less than 30% risk of relapse
9. Known history of known myelodysplastic syndrome

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Metastatic Castrate Resistant Prostate Cancer
Enrollment: 6 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in the proportion of subjects in assessing safety of 225Ac-J591 in those previously treated with PSMA-TRT. | Will be collected at the time of visit 1 through end of study or 100 months
  Proportion of subjects with dose-limiting toxicity (DLT) from treatment cycle 1 to the end of the safety evaluation period at the end of the study. Acceptable safety is determined if no more than 2 (33%) of the subjects in a cohort experience DLT.

SECONDARY OUTCOMES:
Change in the number of subject with Prostate Specific Antigen (PSA) decline following 225Ac-J591 administration | Will be collected at the time of visit 1 through end of study or 100 months
  PSA will be analyzed through blood specimen collection
Change in adverse event rate response | Will be collected at the time of visit 1 through end of study or 100 months
  National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 is used to grade all adverse events
Change in the number of subjects with dose limiting toxicity (DLT) | Will be collected at the time of visit 1 through end of study or 100 months
  DLTs will be measured by the recommended phase I fractionated dose and multiple dose regimens of 225Ac-J591 dose by utilizing the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Change in radiographic response rate | Will be collected at the time of visit 1 through end of study or 100 months
  Radiographic response rate will be captured through radiographic scans such as MRI, CT and bone scans. Response evaluation criteria in solid tumors (RECIST) criteria with Prostate Cancer Working Group 3 (PCWG3) modifications
Change in circulating tumor cells (CTC) response | Will be collected at the time of visit 1 through end of study or 100 months
  CTCs will be analyzed through blood specimen collection via CellSearch methodology lab testing
Change in progression-free survival following re-treatment doses of 225Ac-J591 | Will be collected at the time of visit 1 through end of study or 100 months
Change in Overall Survival Following re-Treatment Doses of 225Ac-J591 | Survival will be collected at the time of visit 1 through end of study or 100 months
  Overall survival will be captured through in-clinic or telephone contact with subjects

CONTACTS AND LOCATIONS:
Overall Officials: Scott Tagawa, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Brooklyn Methodist Hospital - New York Presbyterian, Brooklyn, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No